CLINICAL TRIAL: NCT05456087
Title: Use of Botulinum Toxin in the Treatment of Androgenic Alopecia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zel Skin and Laser Specialists (Other)
Collaborators: Merz Aesthetics Inc. (Industry)
Responsible Party: Principal Investigator, Brian Zelickson, Principal Investigator, Zel Skin and Laser Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEL-IIT5773
Record Dates: First submitted 2022-04-12; First posted 2022-07-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Androgenetic Alopecia
Keywords: Patterned Hair Loss
MeSH Terms: conditions — Alopecia | interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single treatment with Xeomin® (incobotulinumtoxin A) (Experimental): Individual balding scalps will be outlined and mapped to include up to 30 injection sites evenly distributed within the hair loss area. At each site, 5 Units of Xeomin® will be injected with a maximum of 150 Units total per subject. This will be a single, one-time treatment session.
  Interventions: Drug: incobotulinumtoxin A

INTERVENTIONS:
Drug: incobotulinumtoxin A — Up to 150 units of incobotulinumtoxin A will be injected at up to 30 injection sites within the hair loss area
  Other Names: Xeomin

SUMMARY:
The purpose of this study is to evaluate the effect of using a purified botulinum toxin (Xeomin®, Merz, USA), the same injectable used to improve face wrinkles, to treat a specific type of hair loss seen in men and women not associated with scarring or other internal disease called 'pattern hair loss'. This type of hair loss is medically called 'androgenic or androgenetic alopecia'. In men it is typically called 'male pattern baldness' whereas in women it is called 'female pattern baldness' and in both cases is hereditary meaning there will be a history of relatives that describe having the same condition.

DETAILED DESCRIPTION:
Adult volunteers aged 22-55 years presenting with mild to moderate patterned hair loss will be screened for participation. Twenty subjects (10 males and 10 females) meeting the inclusion/exclusion criteria will be recruited to participate. Prior to any injections a global photograph documenting the patterned hair loss will be acquired for each individual utilizing the Canfield global camera system. Each subject will then undergo trichoscopy imaging within the defined treatment area using the Canfield HairMetrix® system. The imaged area is at a higher magnification capable of reliable measurements for hair density (count/cm2), hair shaft diameter, follicular units, among other measurements captured by the software. Individual balding scalps will be outlined and mapped to include up to 30 injection sites evenly distributed within the hair loss area.

At each site, 5 Units of Xeomin® will be injected with a maximum of 150 Units total per subject. This will be a single, one-time treatment session. Consequently, subjects will be contacted by phone or will be asked to come into the clinic for follow up according to a set schedule.

At each follow up visit (monthly) subjects will be asked to report any adverse events. Follow up visits at the clinic will also include photographic documentation, trichoscopy, and investigator and subject subjective reporting of treatment progress.

There will be a total of up to 3 injectors, 1 person taking photographs (including trichoscopy), and 1 investigator assessing treatment outcome.

During this 9 month-long study, subjects cannot utilize other hair loss treatments and must maintain their grooming routine which includes maintaining their hair style.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed by the investigator with mild to moderate degree of hair-pattern loss (androgenic alopecia). Mild to moderate will be defined by investigator assessment of III Vertex-V on the Norwood Scale ( for males) or 3-6 on the Savin Scale (for females).
2. Subjects must be between 22-55 years of age with mild to moderate AGA with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
3. Subjects must agree to maintain the same hair grooming and style routine during study participation.
4. Sexually active females of childbearing potential participating in the study must agree to use a medically-acceptable method of contraception while receiving study product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Exception: Sexually inactive females of childbearing potential are not required to practice a reliable method of contraception and may be enrolled at the investigator's discretion, provided that they understand the possible risks involved in getting pregnant during the study and are counseled to remain sexually inactive for the duration of the study or to practice a reliable method of contraception if becoming sexually active during the study.
5. Subjects must sign a written informed consent.
6. Subjects must sign a photo release form.

Exclusion Criteria:

1. Any systemic treatment for hair loss within the last 6 months including hormonal therapy for peri-menopausal females.
2. Concurrent therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study.
3. Subjects under current treatments in study area with light therapy, microneedling, Platelet-rich Plasma, prostaglandin analogues, ketoconazole, hair transplant or any method deemed unacceptable by the investigator.
4. Any history of drug interaction, such as, aminoglycoside antibiotics, penicillamine, quinine and calcium channel blockers
5. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
6. History of allergic reaction to similar products (Botox® or Dysport®)
7. Albumin sensitivity (allergy to eggs)
8. Subjects with any signs of infection at the injection sites
9. Active cold or sinus infection
10. Any dermatologic or systemic disorder, which in the investigator's opinion, may interfere with the treatment. Examples of such disorders include neuromuscular disorders, hypertrophic scarring, keloidal scarring, bleeding disorders, subjects on immunosuppressive medications, and lupus erythematosus.
11. Subjects who are pregnant, breast feeding or planning a pregnancy during the study period.
12. Subjects who are unwilling or unable to comply with the requirements of the protocol.
13. Participation in another research study (currently or within the last 30 days).
14. All volunteers unwilling to sign the consent forms after being informed of their obligations and risks that they might encounter as a participant in this study.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in hair count per cm2 (number of hairs per follicular unit) | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline hair count per cm2 will be compared to day 30, day 90, day 180 and day 270.
Changes from baseline in sum of hair width per cm2 (total scalp coverage) | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline sum of hair width per cm2 will be compared to day 30, day 90, day 180 and day 270.
Changes from baseline in Terminal:Vellus ratio (number of terminal hairs for every one vellus hair). | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline Terminal:Vellus ratio will be compared to day 30, day 90, day 180 and day 270.
Changes from baseline in Average hairs per follicular unit (average number of hairs within a hair follicle). | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline average hairs per follicular unit will be compared to day 30, day 90, day 180 and day 270.
Changes from baseline in Average hair width (microns) (average thickness of hair in microns). | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline average hair width (microns) will be compared to day 30, day 90, day 180 and day 270.
Changes from baseline in Follicle count per cm2 (number of follicles per square centimeter). | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline follicle count per cm2 will be compared to day 30, day 90, day 180 and day 270.
Mean Inter-follicular distance (mm) (mean distance between follicular units). | Day 30, Day 90, Day 180, and Day 270
  Trichoscopy equipped with Canfield HairMetrix® software system will be performed on the scalp of study participants. The baseline mean inter-follicular distance (mm) will be compared to day 30, day 90, day 180 and day 270.

SECONDARY OUTCOMES:
Change from baseline in balding scalp hair recovery assessed by study investigator | Day 30
  Hair recovery will be assessed by the study investigator on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study investigator | Day 90
  Hair recovery will be assessed by the study investigator on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study investigator | Day 180
  Hair recovery will be assessed by the study investigator on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study investigator | Day 270
  Hair recovery will be assessed by the study investigator on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study participant | Day 30
  Hair recovery will be assessed by the study participant on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study participant | Day 90
  Hair recovery will be assessed by the study participant on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study participant | Day 180
  Hair recovery will be assessed by the study participant on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.
Change from baseline in balding scalp hair recovery assessed by study participant | Day 270
  Hair recovery will be assessed by the study participant on a 4- point scale, where 0 is poor and 3 is excellent. Photographic documentation will be utilized.

CONTACTS AND LOCATIONS:
Locations (1):
- ZelSkin and Laser Specialists, Edina, Minnesota, United States

REFERENCES:
- [Background] Russo PM, Fino E, Mancini C, Mazzetti M, Starace M, Piraccini BM. HrQoL in hair loss-affected patients with alopecia areata, androgenetic alopecia and telogen effluvium: the role of personality traits and psychosocial anxiety. J Eur Acad Dermatol Venereol. 2019 Mar;33(3):608-611. doi: 10.1111/jdv.15327. Epub 2018 Dec 2. PMID 30394586
- [Background] Cash TF. The psychosocial consequences of androgenetic alopecia: a review of the research literature. Br J Dermatol. 1999 Sep;141(3):398-405. doi: 10.1046/j.1365-2133.1999.03030.x. PMID 10583042
- [Background] Bienova M, Kucerova R, Fiuraskova M, Hajduch M, Kolar Z. Androgenetic alopecia and current methods of treatment. Acta Dermatovenerol Alp Pannonica Adriat. 2005 Mar;14(1):5-8. PMID 15818439
- [Background] Norwood OT. Incidence of female androgenetic alopecia (female pattern alopecia). Dermatol Surg. 2001 Jan;27(1):53-4. PMID 11231244
- [Background] Starace M, Orlando G, Alessandrini A, Piraccini BM. Female Androgenetic Alopecia: An Update on Diagnosis and Management. Am J Clin Dermatol. 2020 Feb;21(1):69-84. doi: 10.1007/s40257-019-00479-x. PMID 31677111
- [Background] Inui S, Itami S. Androgen actions on the human hair follicle: perspectives. Exp Dermatol. 2013 Mar;22(3):168-71. doi: 10.1111/exd.12024. Epub 2012 Sep 28. PMID 23016593
- [Background] Ramos PM, Miot HA. Female Pattern Hair Loss: a clinical and pathophysiological review. An Bras Dermatol. 2015 Jul-Aug;90(4):529-43. doi: 10.1590/abd1806-4841.20153370. PMID 26375223
- [Background] Cousen P, Messenger A. Female pattern hair loss in complete androgen insensitivity syndrome. Br J Dermatol. 2010 May;162(5):1135-7. doi: 10.1111/j.1365-2133.2010.09661.x. Epub 2010 Feb 1. PMID 20128792
- [Background] Sinclair R. Winding the clock back on female androgenetic alopecia. Br J Dermatol. 2012 Jun;166(6):1157-8. doi: 10.1111/j.1365-2133.2012.10934.x. No abstract available. PMID 22626036
- [Background] Cotsarelis G, Millar SE. Towards a molecular understanding of hair loss and its treatment. Trends Mol Med. 2001 Jul;7(7):293-301. doi: 10.1016/s1471-4914(01)02027-5. PMID 11425637
- [Background] Goldman BE, Fisher DM, Ringler SL. Transcutaneous PO2 of the scalp in male pattern baldness: a new piece to the puzzle. Plast Reconstr Surg. 1996 May;97(6):1109-16; discussion 1117. doi: 10.1097/00006534-199605000-00003. PMID 8628793
- [Background] Ramos PM, Brianezi G, Martins AC, da Silva MG, Marques ME, Miot HA. Apoptosis in follicles of individuals with female pattern hair loss is associated with perifollicular microinflammation. Int J Cosmet Sci. 2016 Dec;38(6):651-654. doi: 10.1111/ics.12341. Epub 2016 Jun 1. PMID 27163333
- [Background] Garza LA, Liu Y, Yang Z, Alagesan B, Lawson JA, Norberg SM, Loy DE, Zhao T, Blatt HB, Stanton DC, Carrasco L, Ahluwalia G, Fischer SM, FitzGerald GA, Cotsarelis G. Prostaglandin D2 inhibits hair growth and is elevated in bald scalp of men with androgenetic alopecia. Sci Transl Med. 2012 Mar 21;4(126):126ra34. doi: 10.1126/scitranslmed.3003122. PMID 22440736
- [Background] Jaworsky C, Kligman AM, Murphy GF. Characterization of inflammatory infiltrates in male pattern alopecia: implications for pathogenesis. Br J Dermatol. 1992 Sep;127(3):239-46. doi: 10.1111/j.1365-2133.1992.tb00121.x. PMID 1390168
- [Background] Gupta M, Mysore V. Classifications of Patterned Hair Loss: A Review. J Cutan Aesthet Surg. 2016 Jan-Mar;9(1):3-12. doi: 10.4103/0974-2077.178536. PMID 27081243
- [Background] HAMILTON JB. Patterned loss of hair in man; types and incidence. Ann N Y Acad Sci. 1951 Mar;53(3):708-28. doi: 10.1111/j.1749-6632.1951.tb31971.x. No abstract available. PMID 14819896
- [Background] Norwood OT. Male pattern baldness: classification and incidence. South Med J. 1975 Nov;68(11):1359-65. doi: 10.1097/00007611-197511000-00009. PMID 1188424
- [Background] Ludwig E. Classification of the types of androgenetic alopecia (common baldness) occurring in the female sex. Br J Dermatol. 1977 Sep;97(3):247-54. doi: 10.1111/j.1365-2133.1977.tb15179.x. PMID 921894
- [Background] Olsen EA. The midline part: an important physical clue to the clinical diagnosis of androgenetic alopecia in women. J Am Acad Dermatol. 1999 Jan;40(1):106-9. doi: 10.1016/s0190-9622(99)70539-6. No abstract available. PMID 9922024
- [Background] Kasprzak M, Sicinska J, Sinclair R. The Trichoscopy Derived Sinclair Scale: Enhancing visual assessment through quantitative trichoscopy. Australas J Dermatol. 2019 May;60(2):134-136. doi: 10.1111/ajd.12964. Epub 2018 Dec 18. PMID 30565210
- [Background] Sinclair R, Jolley D, Mallari R, Magee J. The reliability of horizontally sectioned scalp biopsies in the diagnosis of chronic diffuse telogen hair loss in women. J Am Acad Dermatol. 2004 Aug;51(2):189-99. doi: 10.1016/s0190-9622(03)00045-8. PMID 15280836
- [Background] Dinh QQ, Sinclair R. Female pattern hair loss: current treatment concepts. Clin Interv Aging. 2007;2(2):189-99. PMID 18044135
- [Background] Afifi L, Maranda EL, Zarei M, Delcanto GM, Falto-Aizpurua L, Kluijfhout WP, Jimenez JJ. Low-level laser therapy as a treatment for androgenetic alopecia. Lasers Surg Med. 2017 Jan;49(1):27-39. doi: 10.1002/lsm.22512. Epub 2016 Apr 25. PMID 27114071
- [Background] Jimenez JJ, Wikramanayake TC, Bergfeld W, Hordinsky M, Hickman JG, Hamblin MR, Schachner LA. Efficacy and safety of a low-level laser device in the treatment of male and female pattern hair loss: a multicenter, randomized, sham device-controlled, double-blind study. Am J Clin Dermatol. 2014 Apr;15(2):115-27. doi: 10.1007/s40257-013-0060-6. PMID 24474647
- [Background] Starace M, Alessandrini A, D'Acunto C, Melandri D, Bruni F, Patrizi A, Piraccini BM. Platelet-rich plasma on female androgenetic alopecia: Tested on 10 patients. J Cosmet Dermatol. 2019 Feb;18(1):59-64. doi: 10.1111/jocd.12550. Epub 2018 Apr 30. PMID 29707872
- [Background] Giordano S, Romeo M, di Summa P, Salval A, Lankinen P. A Meta-analysis On Evidence Of Platelet-rich Plasma for Androgenetic Alopecia. Int J Trichology. 2018 Jan-Feb;10(1):1-10. doi: 10.4103/ijt.ijt_74_16. PMID 29440850
- [Background] Singh S, Neema S, Vasudevan B. A Pilot Study to Evaluate Effectiveness of Botulinum Toxin in Treatment of Androgenetic Alopecia in Males. J Cutan Aesthet Surg. 2017 Jul-Sep;10(3):163-167. doi: 10.4103/JCAS.JCAS_77_17. PMID 29403190
- [Background] Zhou Y, Yu S, Zhao J, Feng X, Zhang M, Zhao Z. Effectiveness and Safety of Botulinum Toxin Type A in the Treatment of Androgenetic Alopecia. Biomed Res Int. 2020 Aug 4;2020:1501893. doi: 10.1155/2020/1501893. eCollection 2020. PMID 32802833
- [Background] Melo DF, Ramos PM, Antelo DAP, Machado CJ, Barcaui CB. Is there a rationale for the use of botulinum toxin in the treatment of Androgenetic Alopecia? J Cosmet Dermatol. 2021 Jul;20(7):2093-2095. doi: 10.1111/jocd.14177. Epub 2021 May 3. No abstract available. PMID 33894053
- [Background] Zhang L, Yu Q, Wang Y, Ma Y, Shi Y, Li X. A small dose of botulinum toxin A is effective for treating androgenetic alopecia in Chinese patients. Dermatol Ther. 2019 Jul;32(4):e12785. doi: 10.1111/dth.12785. Epub 2019 Jan 8. No abstract available. PMID 30566260
- [Background] Unger WP, Unger RH. Hair transplanting: an important but often forgotten treatment for female pattern hair loss. J Am Acad Dermatol. 2003 Nov;49(5):853-60. doi: 10.1016/s0190-9622(03)01568-8. PMID 14576664
- [Background] Kanti V, Messenger A, Dobos G, Reygagne P, Finner A, Blumeyer A, Trakatelli M, Tosti A, Del Marmol V, Piraccini BM, Nast A, Blume-Peytavi U. Evidence-based (S3) guideline for the treatment of androgenetic alopecia in women and in men - short version. J Eur Acad Dermatol Venereol. 2018 Jan;32(1):11-22. doi: 10.1111/jdv.14624. Epub 2017 Nov 27. PMID 29178529
- [Background] Witmanowski H, Blochowiak K. The whole truth about botulinum toxin - a review. Postepy Dermatol Alergol. 2020 Dec;37(6):853-861. doi: 10.5114/ada.2019.82795. Epub 2019 Feb 5. PMID 33603602
- [Background] Martina E, Diotallevi F, Radi G, Campanati A, Offidani A. Therapeutic Use of Botulinum Neurotoxins in Dermatology: Systematic Review. Toxins (Basel). 2021 Feb 5;13(2):120. doi: 10.3390/toxins13020120. PMID 33562846
- [Background] Rakowska A, Slowinska M, Kowalska-Oledzka E, Olszewska M, Rudnicka L. Dermoscopy in female androgenic alopecia: method standardization and diagnostic criteria. Int J Trichology. 2009 Jul;1(2):123-30. doi: 10.4103/0974-7753.58555. PMID 20927234